CLINICAL TRIAL: NCT03678077
Title: 5-year Trend in Cohabitation Status, Academic Achievement and Socio-economic Indicators After Mild Traumatic Brain Injury: a National Register Study
Brief Title: Trends in Cohabitation Status, Academic Achievement and Socio-economic Indicators After Mild Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other); Sygekassernes Helsefond (Other); Aase and Ejnar Danielsens Foundation (Other)
Responsible Party: Principal Investigator, Heidi Jeannet Graff, Phd student, University of Copenhagen
Other Study IDs: mTBI-HJG-2018
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Mild Traumatic Brain Injury; Concussion, Mild; Academic Achievement; Specific Academic or Work Inhibition; Marriage; Marital Status; Income; Education; Socioeconomic Status; Sickness Absence
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mild traumatic brain injury: Patients between 18-60 years, who were hospital admitted, emergency or outpatient treated with mild traumatic brain injury (ICD-10 S06.0). Data were extracted from the Danish national patient register from January 2003 - December 2007.
  Patients who were not resident in Denmark 5 years before and during the inclusion period were excluded (1998-2007).
  Interventions: Other: Mild traumatic brain injury
- Matching controls: Matching controls without concussion of the same age, from the same municipality and of same gender as the included cases. Controls were included during 2003 - 2007. Data were extracted from the population register.
  Controls who were not resident in Denmark 5 years before and during the inclusion period were excluded (1998-2007).

INTERVENTIONS:
Other: Mild traumatic brain injury — This is a register based observational study and does not include interventions. Exposure is mild traumatic brain injury.
  Groups: Mild traumatic brain injury

SUMMARY:
Mild traumatic brain injury (mTBI) accounts for 70-90% of all diagnosed traumatic brain injuries (TBI) affecting approximately 50-300 per 100.000 individuals annually. Persistent post-concussion symptoms are reported in 15-80% of hospital admitted and outpatient treated populations, affecting labour market attachment, academic achievement, income, socio-economic status, social interactions, home management, leisure activities and cohabitation status.

The association between mTBI and long-term trends in cohabitation status, income, academic achievement and socio-economic status has not been thoroughly explored. Previous studies focus on children's academic performance after severe TBI and only few studies include early adulthood and patients with mTBI. Trends in divorce rates are frequently conducted on severe injuries or populations consisting of veterans. Additionally, all studies have failed to apply a national register based design.

Aim The aim of the study is to examine the long-term associations between mTBI and trends in cohabitation status, academic achievement and socio-economic status between pre-injury rates and observed rates at 5 years post-injury. The hypothesis was that by 5 years mTBI would be associated with increased odds of marital breakdown, decreasing academic achievement, decreasing income, decreasing socio-economic status compared to the general population in Denmark.

Methods:

The study is a national register based cohort study with 5 years follow-up of patients with mild traumatic brain injury from 2008 - 2012 in Denmark.

Population:

Patients between 18-60 years diagnosed with concussion (ICD-10 S06.0) were extracted from the Danish National Patient Register between (2003-2007). Patients with major neurological injuries and previous concussions at the index date and 5 years before the index date (1998-2007) were excluded. Patients who were not resident in Denmark 5 years before and during the inclusion period were also excluded (1998-2007).

Data will be retrieved from several national databases, including: the Danish national patient register, Danish Civil Registration System (CRS), the Danish Education Registers, the Income Statistics Register and the Employment Classification Module (AKM).

One control of the general population were matched for each case on sex, age and municipality.

Outcome measures are: Cohabitation status, Education, income and socio-economic status.

ELIGIBILITY:
Inclusion Criteria:

* Concussion (ICD-10 S06.0) (primary diagnosis)(2003-2007)

Exclusion Criteria:

* Major neurological injuries and previous concussions (1998-2007)
* Not resident in Denmark (1998-2007)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Hospital admitted, emergency or outpatient treated patients between 18-60 years diagnosed with concussion (ICD-10 S06.0) are extracted from the Danish National Patient Registre between (2003-2007).
Sampling Method: Probability Sample
Enrollment: 45777 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Cohabitation status | 5 years follow-up (2008-2012)
  Data comprise four definitions of married couples, registered partnerships, couples living in consensual union, cohabiting couple or being single. Data were consolidated into married/cohabiting couple or single status.

SECONDARY OUTCOMES:
Education | 5 years follow-up (2008-2012)
  The highest completed qualifying education, given at the index date was used as a measure of academic achievement. Data were categorized into high education vs. low education. Low education encompasses basic schooling, high school, trade and craft educations and high educations encompass short education, medium length education, bachelor's degree, university degrees and Ph.D.
Income | 5 years follow-up (2008-2012)
  To describe long-term trends in income, we analyze data on personal gross income including revenue and social transfer income and categorized data into two income groups: Low annually income (<200.000 DKK). and high annually income (>200.000 DKK).
Socioeconomic status | 5 years follow-up (2008-2012)
  Based on occupation and income, socio-economic status determines whether the person is employed, unemployed or outside the labour force. To measure how mTBI influences socioeconomic status (employment status) regarding occupation and labour market attachment, data were categorized into (1) Self-employed/leaders/managers vs. wage earners/enrolled in education/not economically active and (2) Gainfully employed vs. not economically active.

CONTACTS AND LOCATIONS:
Overall Officials: Hana M Rytter, Study Director — Department of Psychology
Locations (1):
- Department of Psychology, University of Copenhagen, Copenhagen, DK, Denmark

IPD SHARING:
Plan to Share IPD: No